CLINICAL TRIAL: NCT02269072
Title: Testosterone Regulation of the Natriuretic Peptide System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Director, Neuroendocrine Research Program in Women's Health, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2014P00
Record Dates: First submitted 2014-10-15; First posted 2014-10-20 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
Keywords: Natriuretic Peptide
MeSH Terms: conditions — Hypertension | interventions — Testosterone; Natriuretic Peptide, Brain; Leuprolide; Anastrozole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Active Comparator): Testosterone cream applied daily
  Interventions: Drug: Testosterone; Drug: Nesiritide; Drug: Leuprolide; Drug: Anastrozole
- Placebo (Placebo Comparator): Identical placebo cream applied daily
  Interventions: Drug: Nesiritide; Drug: Leuprolide; Drug: Anastrozole; Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — Testosterone cream applied daily for two weeks
  Arms: Testosterone
Drug: Nesiritide — Administered IV once during the study
Drug: Leuprolide — Administered twice during the study by injection
Drug: Anastrozole — Daily pill for 8 weeks
Drug: Placebo — Inert cream otherwise identical to testosterone cream applied daily for two weeks
  Arms: Placebo

SUMMARY:
The proposed study is a physiologic investigation of the effects of testosterone on the natriuretic peptide system. The hypotheses of the study are that testosterone administration will decrease natriuretic peptide levels and salt excretion. The entire protocol is 8 weeks in duration.

ELIGIBILITY:
Inclusion Criteria:

* Men: aged 18 to 40 years, normal testosterone and free testosterone levels, no history of hypertension, and BMI between 18.5 and 25.
* Women: aged 18 to 40 years old, regular menstrual periods, negative pregnancy test, no oral contraceptives for ≥ 3 mos, no history of hypertension, BMI between 18.5 and 25.

Exclusion Criteria:

* Antihypertensives, diuretics or insulin, diabetes mellitus, prior cardiovascular, abnormal liver or renal disease, history of cancer, atrial fibrillation, or abnormal sodium or potassium level.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Atrial natriuretic peptide levels | 8 weeks

SECONDARY OUTCOMES:
Urinary salt excretion | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen K Miller, MD, Principal Investigator — Massachusetts General Hospital